CLINICAL TRIAL: NCT01235923
Title: A Randomized, Masked Study of Weekly Erythropoietin Dosing in Preterm Infants
Brief Title: Randomized Study of Weekly Erythropoietin Dosing in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-380; M01RR000997 (NIH)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2012-06

CONDITIONS: Preterm Infants
Keywords: anemia; transfusions; erythropoiesis; neonate; preterm
MeSH Terms: conditions — Anemia; Premature Birth | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- three times weekly Epo (Active Comparator): Epo 400 units/kg three times weekly given subcutaneously for 4 weeks
  Interventions: Drug: three times weekly Epo
- weekly Epo (Active Comparator): 1,200 units/kg given once a week subcutaneously for 4 weeks
  Interventions: Drug: weekly Epo

INTERVENTIONS:
Drug: three times weekly Epo — Epo 400 units/kg administered subcutaneously three times per week for a total of 4 weeks
  Other Names: Epoetin alfa; Procrit
  Arms: three times weekly Epo
Drug: weekly Epo — Epo 1,200 units/kg administered subcutaneously once a week for a total of 4 weeks
  Other Names: Epoetin alfa; Procrit
  Arms: weekly Epo

SUMMARY:
Preterm infants are a risk for multiple transfusions, and the administration of human recombinant erythropoietin (Epo) has been shown to decrease transfusion requirements. Dosing usually occurs three times a week, but extended dosing schedules have been successful in adults. The investigators assessed weekly Epo dosing in preterm infants compared to standard three times weekly dosing.

DETAILED DESCRIPTION:
Erythropoietin (Epo) increases and maintains hematocrit using once weekly dosing in adults with anemia due to end stage renal disease. Epo is used in preterm infants to treat the anemia of prematurity, but has not been studied using once weekly dosing. We compared reticulocyte responses of once weekly Epo dosing with thrice weekly dosing in preterm infants.

Infants ≤1,500 grams and ≥7 days of age were randomized to once weekly Epo, 1,200 units/kg/dose, or thrice weekly Epo, 400 units/kg/dose, subcutaneously for 4 weeks, along with iron and vitamin supplementation. Complete blood counts, absolute reticulocyte counts (ARC), transfusions, phlebotomy losses, and adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

* < or = 1,500 grams
* < or = 32 weeks gestation
* > or = 7 days of age
* informed consent obtained

Exclusion Criteria:

* hemolytic disease
* hypertension
* seizures
* thromboses
* major malformation

Ages: 7 Days to 100 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin K Ohls, MD, Principal Investigator — University of New Mexico
Locations (1):
- UNM NICU, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants ≤1,500 grams and ≥7 days of age hospitalized in the NICU at UNM between 4/06 and 3/09 were randomized to once weekly Epo, 1,200 units/kg/dose, or thrice weekly Epo, 400 units/kg/dose, subcutaneously for 4 weeks, along with iron and vitamin supplementation.
Groups:
- Weekly Epo: Epo 1,200 units/kg given once a week subcutaneously for 4 weeks
Period: Overall Study
Arm/Group | Three Times Weekly Epo | Weekly Epo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Three Times Weekly Epo | Weekly Epo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Mean (Standard Deviation); unit: days] | 15 (4) | 18 (3) | 17 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Baseline Retic Count
Description: retic count measured at study entry
Time Frame: baseline
Population: All study subjects had baseline retic count measured.
Measure: Mean (Standard Error); unit: x1000 cells/microliter
Arm/Group | Weekly Epo | Three Times a Week Epo
Number analyzed (Participants) | 10 | 10
x1000 cells/microliter | 122 (12) | 140 (24)

2. Primary Outcome: Reticulocyte Count
Description: reticulocyte count at 4 weeks (end of study)
Time Frame: 4 weeks
Population: Power analysis based on difference in mean retic count (baseline versus 4 weeks) of 75 (standard deviation 50), alpha 0.05, 80% power.
Measure: Mean (Standard Error); unit: cells x 1000/microliter
Arm/Group | Weekly Epo | Three Times a Week Epo
Number analyzed (Participants) | 10 | 10
cells x 1000/microliter | 275 (70) | 268 (34)

ADVERSE EVENTS:
Arm/Group | Weekly Epo | Three Times Weekly Epo
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly Epo (N=10) | Three Times Weekly Epo (N=10)
Death (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly Epo (N=10) | Three Times Weekly Epo (N=10)
bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) — oxygen requirement at 36 weeks adjusted age
interventricular hemorrhage greater than grade 2 (Nervous system disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
pilot study with only 20 infants evaluated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes